CLINICAL TRIAL: NCT03127475
Title: Neurophysiological Dissection and Intervention of Freezing of Gait in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The chief, Department of Neurology, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH105-REC1-004
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Parkinson's Disease With Freezing of Gait
Keywords: Parkinson's disease; freezing of gait; electrophysiology; magnetic resonance image; direct current stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): Device: Transcranial direct current stimulation In tDCS,the anodal pad was tapped over the primary motor cortex and the cathode pad was adhered of the contralateral frontal region. A constant current of 2.0 mA will be apply for up to 20 min, with a linear fade in /fade out of 10 s in anodal and cathodal conditions resulting in a current density of 0.8A/M2 which is 177 times below the lesion effect of tDCS in the rats study(142.9A/m2)
  Interventions: Device: Transcranial direct current stimulation
- sham tDCS (Sham Comparator): Device: Sham tDCS Sham stimulation will be 30s stimulation with ramp up and ramp off for 10s at 2.0 mA.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — A consecutive 5-days course of tDCS will be delivered. In treatment group, true stimulation will be administrated and sham stimulation will be delivered in control group.

SUMMARY:
Different conditions of gait ignition freezing, spontaneous freezing during walking and turning freezing on encountering obstacle will be investigated in fMRI study to examine whether different regions of brain will be involved under different conditions of freezing. We hypothesize that anterior cortical regions will engage in gait ignition failure, deep locomotion regions will be responsible for spontaneous freezing and schema regions will be involved in the generation of turning freezing on seeing the barrier. In the third part of the project, we will deliver a 5-day session of transcranial direct current stimulation (tDCS) to the motor cortex of the FOG patients to examine whether the intervention will benefit the patients. Based on the signal source findings, we will investigate whether the possible tDCS beneficial effect will be different or similar in patients with different electric sources. In addition, how long the possible beneficial effect of tDCS can be consolidated after the 5-day course of stimulation is crucial and requires to be elucidated under the research project. We aim to peep the myth of FOG in PD by the multi-modality approach and hope the study will benefit the long suffering patients.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of freezing of gait will be made by the following criteria:

1. Without video:Is there any feeling that your feet are transiently glued to the floor while trying to initiate walking, making a turn or when walking through narrow spaces or in crowded places? (Sometimes it can be accompanied with trembling of the legs and small shuffling steps.)
2. Additional instructions with video:We will watch a short video together to see the many ways in which freezing can occur. Also, look carefully for how long these episodes last, as you can expect some questions on this later.
3. Patient is diagnosed to have freezing of gait if "I have experienced such a feeling or episode over the past month" was answered.

Exclusion Criteria:

1. Impairment of cognition that leads unable to fully cooperate with the oral commands during examinations.
2. Moderate to severe medical disorders such as functional III or above congestive heart failure, or cancer with distant metastasis etc.
3. Hoehn and Yahr stage 5.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in laboratory gait analysis after the tDCS session | baseline to week 4
  Variables in gait analysis:1.Gait initiation, 2.Level walking, 3.Turning, 4.Gait termination

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) after the tDCS session | baseline to week 4

OTHER OUTCOMES:
Change in the 39-item Parkinson's Disease Questionnaire (PDQ-39) after the tDCS session | baseline to week 4
Change in non-motor symptom assessment scale for Parkinson's Disease after the tDCS | baseline to week 4
Change in Fall assessment test after the tDCS session | baseline to week 4
Change in new freezing of gait questionnaire(NFOG-Q) after the tDCS session | baseline to week 4
Change in Tinetti's Mobility Index after the tDCS session | baseline to week 4

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided